CLINICAL TRIAL: NCT01777672
Title: Effect of Afferent Oropharyngeal Pharmacological and Electrical Stimulation on Swallow Response and on Activation of Human Cortex in Stroke Patients With Oropharyngeal Dysphagia (OD). A Randomized Controlled Trial.
Brief Title: Effect of Afferent Oropharyngeal Pharmacological and Electrical Stimulation on Swallow Response and on Activation of Human Cortex in Stroke Patients With Oropharyngeal Dysphagia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital de Mataró (Other)
Responsible Party: Principal Investigator, Pere Clave, MD, PhD, Hospital de Mataró
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Marató-11
Record Dates: First submitted 2013-01-21; First posted 2013-01-29 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Dysphagia; Aspiration; Stroke
MeSH Terms: conditions — Deglutition Disorders; Stroke | interventions — Diet; Electrodes; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (4):
- Dietary and oral hygiene recommendations (Active Comparator): Patients in this group will receive recommendations from their healthcare providers about bolus volume and viscosity adaptation for fluids, dietary and nutritional adjustments (liquids and solids) of bolus volume and viscosity/texture. Before leaving each hospital they will also learn basic rehabilitation strategies for OD including swallow postures, compensatory manoeuvres and oropharyngeal rehabilitation exercises and oral hygiene to follow at home.
  Interventions: Behavioral: Dietary and oral hygiene recommendations
- oral TRPV1 agonist (Experimental): Patients will receive the same recommendations as the control group and also recommendation for the administration of a TRPV1 agonist (natural capsaicin) supplement (5 mL bolus before each meal), 3 meals/day, 5 days/week for 2 consecutive weeks.
  Interventions: Behavioral: Dietary and oral hygiene recommendations; Dietary Supplement: oral TRPV1 agonist
- pharyngeal electrical stimulation (Experimental): Treatment in this group will also include the same measures as in the control group, plus neuron stimulation treatment of 1 session / day of pharyngeal electrical stimulation of 10 min duration, 3 days/week during one week, done at the same center.
  Interventions: Behavioral: Dietary and oral hygiene recommendations; Device: pharyngeal electrical stimulation
- transcutaneous electrical stimulation (Experimental): Treatment in this group will be the same as the control group plus trans-cutaneous electrical stimuli will be applied 5 seconds every minute during 1 hour daily session, 5 days/week during 2 consecutive weeks at the same centre.
  Interventions: Behavioral: Dietary and oral hygiene recommendations; Device: transcutaneous electrical stimulation

INTERVENTIONS:
Behavioral: Dietary and oral hygiene recommendations
Dietary Supplement: oral TRPV1 agonist — Patients will receive the administration of a TRPV1 agonist (natural capsaicin) supplement before each meal, 3 meals/day, 5 days/week for 2 consecutive weeks. The TRPV1 agonist will be provided by the pharmacy of the center.
  Arms: oral TRPV1 agonist
Device: pharyngeal electrical stimulation — Includes neuron stimulation treatment of 1 session / day of pharyngeal electrical stimulation of 10 min duration, 3 days/week during 1 week, done at the same center.
  Other Names: Electrodes (Gaeltec, Ltd, Dunvegan, Isle of Skye, UK.; Electrical stimulator (Grass Instruments Co, USA)
  Arms: pharyngeal electrical stimulation
Device: transcutaneous electrical stimulation — Trans-cutaneous electrical stimuli will be applied 5 seconds every minute during 1 hour daily session, 5 days/week during 2 consecutive weeks at the same centre.
  Other Names: Intelect VitalStim, Chattanooga, USA)
  Arms: transcutaneous electrical stimulation

SUMMARY:
Oropharyngeal dysphagia (OD) is a major complaint among many patients with stroke and causes severe complications. There is no specific treatment for these patients. Impaired swallow response is caused by a delay in the timing of oropharyngeal reconfiguration with delayed airway protection. Swallow response is initiated by sensory afferent fibers in the oropharynx and cerebral cortex reaching the central swallowing pattern generator (CPG) in the medulla oblongata and brainstem motor nuclei. Hypothesis: Stimulation of pharyngeal sensory afferent fibers through TRPV1 receptors and electrical stimuli might enhance the stimulation of the CPG and speed the swallow response. Long-term treatment of OD will improve clinical outcome of stroke patients. Aim: To assess the effect of TRPV1 agonists (capsaicin) and that of sensorial pharyngeal electrical stimulation (intrapharyngeal and transcutaneous) on VFS signs and swallow response at 3, 6 and 12 months after treatment in stroke patients with established OD. To compare the clinical effect of classical rehabilitation strategies with that of these new afferent sensorial neurostimulation strategies in terms of nutritional status parameters, incidence of aspiration pneumonia and/or low respiratory tract infection, quality of life, and mortality. Methods: Clinical screening of OD with the volume-viscosity swallow test and assessment by VFS and quantitative measurements of swallow response. Randomized controlled trial assessing the effect of standard rehabilitation with that of afferent sensorial neurostimulation strategies.

ELIGIBILITY:
Inclusion Criteria:

- Person with persistent clinical signs or symptoms of OD according to V-VST and confirmed with VFS (PA scale level 3 or more) secondary to a stroke episode in the last 3 months.

Exclusion Criteria:

* Patient unconscious or in a coma
* Patients diagnosed with transitory ischemic accident
* life expectancy less than 3 months
* neurodegenerative disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-10; Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy and safety of new neuron-stimulation treatments for OD in patients with stroke and to explore their mechanism of action. | 12 months
  The efficacy of each treatment will be assessed by VFS in each patient after the treatment and at the end of the follow-up period, considering Rosenbek scale and measures of oropharyngeal swallow response including oropharyngeal reconfiguration, timing and extent of hyoid motion and bolus propulsion force of the tongue. Clinical outcome also evaluated are episodes of aspiration pneumonia and low respiratory tract infections, nutritional status, complications and clinical symptoms experimented during one year of follow-up and mortality rates and cause of death.
  Participating clinicians will be instructed to register and describe all serious adverse events (SAE) occurred during the study and report them on a specific form within 24 hours. The guidelines for SAE reporting to the Ethical Committee and competent authorities will be followed.

SECONDARY OUTCOMES:
To determine the prevalence of OD and its complications in stroke patients over one year. | 12 months

OTHER OUTCOMES:
To assess and compare one year health resource consumption between all study treatment groups. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pere Pere, Doctor, Principal Investigator — Hospital de Mataró, Gastrointestinal Physiology Laboratory
Locations (1):
- Hospital de Mataró, Mataró, Barcelona, Spain